CLINICAL TRIAL: NCT00488644
Title: Combined Levothyroxine/Liothyronine Supplementation in Hypothyroid Patients With Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0804
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Hypothyroidism; Brain Tumor
Keywords: Hypothyroidism; Brain Tumor; Levothyroxine; Liothyronine; Synthroid; Cytomel
MeSH Terms: conditions — Hypothyroidism; Brain Neoplasms | interventions — Thyroxine; Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levothyroxine + Liothyronine (Experimental): Levothyroxine 75 mcg by mouth (PO) Daily for 8 Weeks + Liothyronine 15 mcg PO Daily for 8 Weeks
  Interventions: Drug: Levothyroxine; Drug: Liothyronine

INTERVENTIONS:
Drug: Levothyroxine — 75 mcg by mouth (PO) Daily for 8 Weeks
  Other Names: Synthroid
Drug: Liothyronine — 15 mcg PO Daily for 8 Weeks
  Other Names: Cytomel

SUMMARY:
Primary Objectives:

1. Assess whether combined treatment with Levothyroxine and Liothyronine improves learning and memory.
2. Explore the relationship between T3 treatment and other domains of cognitive function, quality of life, and mood.

DETAILED DESCRIPTION:
Hypothyroidism causes the body to not be able to produce enough thyroid hormones. Levothyroxine and liothyronine are synthetic (man-made) hormones that may help treat hypothyroidism by increasing the metabolism (activity) of cells of all tissues in the body. The combination treatment, given to patients with hypothyroidism, may help improve normal body and brain functioning.

Levothyroxine is a man-made type of hormone that is made and released by the thyroid gland (thyroxine [T4]). Liothyronine is also a man-made type of hormone, but it is made by the thyroid gland (triiodothyronine [T3]). Both levothyroxine and liothyronine effect different functions in the body that help regulate (control) the activity and amount of energy that cells use.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have your complete medical history recorded. You will have a neuropsychological evaluation (a series of tests that evaluate how well your brain is performing). This evaluation includes an interview, and tests will be performed to check your memory, language, and thinking abilities. You will have a neurological exam performed, which will include measurement of your weight, height, and performance status (how well you are able to perform daily activities). This will be done within 14 days before the start of this study.

You will have blood collected (about 2 tablespoons) for routine laboratory tests (free T4, total T3) for patients with hypothyroidism. You will also be given 4 questionnaires to fill out that will ask about your general QoL and changes in your mood. These questionnaires will take about 20 minutes total to complete.

If you are found to be eligible to take part in this study, you will receive your standard dose of levothyroxine (after you have your blood collected for laboratory tests and physical measurements taken) by mouth. You will receive liothyronine by mouth on Day 1 of this study and then have a neuro-cognitive test ( that evaluates how well your brain is performing). The dose of liothyronine you receive will depend on the dose of levothyroxine that you are already on.

Approximately 4 weeks after you start on the treatment, you will be called by a research data coordinator or research nurse who will ask you questions about any symptoms of hyperthyroidism that you may be having. This is in case your dose of liothyronine is too high and may need to be adjusted.

You will be receiving levothyroxine and liothyronine for up to 8 weeks. However, you will be taken off this study, if your disease gets worse or you experience any intolerable side effects.

You will be asked to return again to the hospital 8 weeks after your first visit for an end-of-study visit. You will have another neuropsychological evaluation performed. Blood (around 2 tablespoons) will again be collected to test the levels of free T4 and total T3 in your body. You will also have your physical measurements taken. You will receive another standard dose of levothyroxine. You will have another neurocognitive test performed, and you will be given 4 more questionnaires to evaluate your QoL and any changes in your mood. The questionnaires will take about 20 minutes total to complete.

Your participation in this study will be over after your end-of-study visit.

This is an investigational study. Liothyronine and levothyroxine each are approved by the FDA for hypothyroidism and are commercially available. However, the use of these drugs in combination is experimental. Up to 26 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have the diagnosis of hypothyroidism.
* Patients must be already on thyroid hormone replacement.
* Patients must be greater than or equal to 18 years old.
* Patients must have a diagnosis of a primary or secondary brain tumor and must have received prior radiation.
* Patients must have a life expectancy of at least 6 months.

Exclusion Criteria:

* Previously established dementing illness.
* Other medical conditions known to cause dementia.
* Significant psychiatric illness.
* Uncontrolled seizures.
* Acute or chronic pulmonary disease.
* Active severe infections.
* Signs or symptoms of coronary artery disease.
* History of congenital hypothyroidism, hyperthyroidism, thyroidectomy, 131I-therapy, or thyroid cancer.
* Paroxysmal supraventricular tachycardia, or any serious unstable medical condition.
* Inability to read and write in English.
* Patients must not be taking any medications that interfere with thyroid hormone metabolism (Beta-Adrenergic Blocking Agents, Antiarrhythmic drugs, Antipsychotic Agents, Tricyclic Antidepressants, Amiodarone, Iodine, Lithium, and Alpha-Interferon).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Levin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 16, 2006 to September 10, 2008. All participants recruited at The University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Levothyroxine + Liothyronine
Started | 12
Completed | 10
Not Completed | 2
Not completed — Not Eligible | 1
Not completed — Not Evaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Levothyroxine + Liothyronine
Number analyzed (Participants) | 12
Age Continuous [Median (Full Range); unit: years] | 44 [33 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating Improvement With Impaired Neuro-cognitive Function (NCF) Based on Results of a Series Neuro-cognitive Exams Administered at Baseline and 8 Weeks After Liothyronine Therapy
Description: At baseline, each participant's scores for standardized/widely-used NCF exams are recorded (recalled words/objects/sequence repetition/etc per tests listed below). After 8 weeks liothyronine therapy, participants are tested again and scores compared to baseline scores. If the participant recalls more numbers/objects/sequence repetition faster/etc., than previous scores, this constitutes an improvement in NCF function for that individual. Scores are not compared to other participants. NCF tests: Memory by RAVLT (Rey Auditory Verbal Learning Test), scored by the number of words correctly recalled at different timepoints; Attention by Digit Span Exam (accurately repeating a sequence of numbers just spoken); Processing speed by Digit Symbol Exam (accurately matching numbers with associated symbols) Executive function by Trail Making Tests and Controlled Oral Word Association; Motor dexterity evaluated by correctly placing pegs in pegboards in a specified time.
Time Frame: At baseline and after 8 weeks of treatment
Measure: Number; unit: participants
Groups:
- 8 Weeks Post Therapy: Levothyroxine 75 mcg by mouth (PO) Daily for 8 Weeks + Liothyronine 15 mcg PO Daily for 8 Weeks.
Arm/Group | 8 Weeks Post Therapy
Number analyzed (Participants) | 10
participants
  Memory function (RAVLT) | 0
  Attention (digit span) | 0
  Processing speed (digit symbol) | 1
  Executive function (trail making) | 3
  Motor dexterity (pegs/pegboard) | 1

ADVERSE EVENTS:
Time Frame: 21 months
Arm/Group | Levothyroxine + Liothyronine
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine + Liothyronine (N=12)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Puritis/Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Metabolic/Lab (Metabolism and nutrition disorders) | 1 (1)
Mood Alteration (Anxiety) (Psychiatric disorders) | 1 (1)
Mood Alteration (Depression) (Psychiatric disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No